CLINICAL TRIAL: NCT03036111
Title: Effect of Trimebutine on Postoperative Pain After Milligan-Morgan Hemorrhoidectomy: A Randomized Controlled Trial
Brief Title: Effect of Topical Trimebutine on Pain After Hemorrhoidectomy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Unavailability of Triembutine maleate
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansourau20172
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-01

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Trimebutine; Hemorrhoidectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemorrhoidectomy (Sham Comparator): Patients will undergo Millgan-Morgan hemorrhoidectomy as classically described before
  Interventions: Procedure: Hemorrhoidectomy
- trimebutine (Active Comparator): Patients will undergo Millgan-Morgan hemorrhoidectomy then triembutine suppository will be inserted in the anal canal intraoperatively and then every six hours for 24 hours.
  Interventions: Drug: Trimebutine; Procedure: Hemorrhoidectomy

INTERVENTIONS:
Drug: Trimebutine — Trimebutine suppository will be inserted in the anal canal on completion of hemorrhoidectomy then at six and 12 hours postoperatively.
  Other Names: Gastreg suppository
  Arms: trimebutine
Procedure: Hemorrhoidectomy — Patients will undergo classic Milliagn-Morgan hemorrhoidectomy

SUMMARY:
Trimebutine acts through smooth muscle relaxation. It is presumed that the topical application of trimebutine after hemorrhoidectomy may help relieve pain after the procedure by relaxing the internal anal sphincter spasm.

DETAILED DESCRIPTION:
A randomized trial will be carried out to investigate the effect of trimebutine on pain after Milligan-Morgan hemorrhoidectomy. Trimebutine relaxes the internal anal sphincter spasm which usually occurs after excisional hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aging between 18-70 years with grade III/VI internal hemorrhoids will be included

Exclusion Criteria:

* Patients with grade I/II internal hemorrhoids or external hemorrhoids.
* Patients with associated anorectal pathology such as anal fissure, anal fistula, rectal prolapse, neoplasm, solitary rectal ulcer, and inflammatory bowel diseases.\
* Patients with recurrent hemorrhoids after previous surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment assessed using visual analogue score from 0-10 | Pain will be assessed at 12 hours after the procedure
  Anal pain will be assessed using visual analogue score from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No